CLINICAL TRIAL: NCT05686681
Title: Improving Social Connectedness in Homebound Older Adults by Integrating a Brief Evidence-Based Telehealth Intervention Into Area Agency on Aging Services
Brief Title: Connect ME: Improving Social Connectedness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Renee.L.Pepin, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02001734
Record Dates: First submitted 2022-12-22; First posted 2023-01-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Social Connectedness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brief Behavioral Activation for Improving Social Connectedness (Experimental): Active, 6 session Brief Behavioral Activation for Improving Social Connectedness
  Interventions: Behavioral: Brief Behavioral Activation for Improving Social Connectedness

INTERVENTIONS:
Behavioral: Brief Behavioral Activation for Improving Social Connectedness — Brief Behavioral Activation for Improving Social Connectedness (BBAISC): BBAISC was developed to address social connectedness. Grounded in Behavioral Activation (Lejuez et al., 2011), BBAISC is a structured, 6-session skill-building intervention that has 4 key elements (Pepin et al., 2020):
  1. Psychoeducation: Psychoeducation focused on homebound status, social connectedness, and associated changes in behavior.
  2. Behavioral Activation intervention rationale: Framing how changing behavior can positively impact social connectedness (i.e., improve social connectedness and reduce loneliness).
  3. Exploration of life areas, values, and activities: Focused on identifying life areas and values most relevant to the participant. Then, these values are used to generate activities that are aligned with those values.
  4. Activity monitoring and planning: Participants are encouraged to schedule and organize their day based on what is important rather than their current mood or feeling state.

SUMMARY:
To assess the reach and effectiveness of a behavioral activation intervention for older adults experiencing low social connectedness by Area Agency on Aging Staff.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (age>60) will be enrolled because they are the target population served by the home-delivered meals program and the target sample for this study.

Exclusion Criteria:

* Clinically significant depression (Patient Health Questionnaire; PHQ-9 ≥ 10) or active suicide risk (Columbia Suicide Severity Rating Scale; C-SSRS), or Cognitive Impairment (Blessed Orientation-Memory-Concentration Test>9)
* Clients who score 1 or greater on question 9 of the PHQ-9 will be further assessed for suicide risk using the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Clients will meet exclusion criteria for a positive response to any item
* We will exclude older adults with uncorrectable hearing or vision impairment rendering them unable to use the tele-conferencing equipment.
* Those who cannot speak English and have impaired decision-making capacity
* Adults unable to consent will be excluded
* Individuals who are not yet adults (infants, children, teenagers) will be excluded
* Pregnant women will be excluded
* Prisoners will be excluded

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Social Connectedness A, Baseline | before the intervention
  10-item Duke Social Support Index (DSSI)
Social Connectedness A, Change from Baseline to Post Intervention | immediately following the intervention
  10-item Duke Social Support Index (DSSI)
Social Connectedness A, Change from Post Intervention to Follow Up | 12 weeks post intervention
  10-item Duke Social Support Index (DSSI)
Social Connectedness B, Baseline | before the intervention
  8-item PROMIS Social Isolation Scale
Social Connectedness B, Change from Baseline to Post Intervention | immediately following the intervention
  8-item PROMIS Social Isolation Scale
Social Connectedness B, Change from Post Intervention to Follow Up | 12 weeks post-intervention
  8-item PROMIS Social Isolation Scale

SECONDARY OUTCOMES:
Intervention Reach | 12 Months
  Reach will be determined by the proportion of eligible agency clients who agree participate in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Renée L Pepin, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No